CLINICAL TRIAL: NCT05494892
Title: Entwicklung Einer Forschungsagenda Für Die Reha-Forschung in Der Österreichischen Pensionsversicherungsanstalt (PVA) [Development of a Research Agenda for Rehabilitation Research in the Austrian Pension Insurance Institution (PVA)]
Brief Title: Development of a Research Agenda for Rehabilitation Research
Status: Completed | Type: Observational
Sponsor: Pensionsversicherungsanstalt (Other)
Responsible Party: Sponsor
Other Study IDs: 0004 Masterplan Reha-Forschung
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-01

CONDITIONS: Research Agenda; Conditions Influencing Health Status
Keywords: Research Agenda; Applied Rehabilitation Research; Expert Survey; Expert Interviews; Delphi Survey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
An internal research department was established in the course of an organisational reform of the Pension Insurance Institution in 2020 for the evidence-based development of its own services in Austria. The focus is on the transfer of findings into practice and the scientific community. As part of an initial assessment of the current situation, an organisation-specific research agenda is being systematically developed.

The project design is based on a multi-perspective and multi-method approach. After obtaining experts' opinions (interview) from different settings and areas, a consensus on necessary fields of action will be worked out after synthesising the results via a Delphi survey.

ELIGIBILITY:
Inclusion Criteria:

* Researchers who conduct scientific research in the field of rehabilitation in Austria, Germany and Switzerland
* People working in rehabilitation facilities (in therapy or administration) in Austria, Germany and Switzerland

Exclusion Criteria:

* Failure to obtain the declaration of consent

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: International and Austrian experts from science and research related to rehabilitation, cooperation partners, representatives of the rehabilitation facilities of the PVA, as well as decision-makers of the PVA were included.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Identification of priorities in applied rehabilitation research | April 2021 - November 2021
  Semi-structured, guideline-based expert interviews with representatives of different stakeholder groups from Austria, Germany and Switzerland are conducted.
  The transcribed interviews are extracted and evaluated within the framework of a qualitative content analysis according to Gläser & Laudel (2010).
  Additionally, based on a scoping review on international research priorities and research agendas in the context of rehabilitation, potentially not considered content will be identified and supplemented.
Weighting of the identified priorities in research | May 2023 - August 2023
  A Delphi survey is conducted with (1) the interview partners and rehabilitation researchers and (2) other representatives of different stakeholder groups from Austria, Germany and Switzerland to evaluate the priorities of the developed research field. The experts are consulted repeatedly until a consensus can be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Stöhr, Mag., Principal Investigator — Pensionsversicherungsanstalt
Locations (1):
- Pensionsversicherungsanstalt, Vienna, Vienna, Austria